CLINICAL TRIAL: NCT03639506
Title: A Pilot Study of the Effect of Autologous Mitochondria Transplantation in Assisted Reproductive Technology Clinical Outcome.
Brief Title: Clinical Application of Autologous Mitochondria Transplantation for Improving Oocyte Quality.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, doctor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: newivf20180817
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Repetition Failure
Keywords: repetition failure; autologous mitochondria transplantation; embryo quality; live birth rate
MeSH Terms: interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- autologous mitochondria transplantation (Experimental): inject autologous mitochondria from bone marrow mesenchymal stem cells into oocyte as well as intracytoplasmic sperm injection (ICSI)
  Interventions: Procedure: autologous mitochondria transplantation; Combination Product: autologous mitochondria from bone marrow mesenchymal stem cells into oocyte as well as intracytoplasmic sperm injection (ICSI)
- ICSI (Active Comparator): only has intracytoplasmic sperm injection (ICSI)
  Interventions: Drug: intracytoplasmic sperm injection (ICSI)

INTERVENTIONS:
Procedure: autologous mitochondria transplantation — inject autologous mitochondria from bone marrow mesenchymal stem cells into oocyte
  Arms: autologous mitochondria transplantation
Combination Product: autologous mitochondria from bone marrow mesenchymal stem cells into oocyte as well as intracytoplasmic sperm injection (ICSI) — autologous mitochondria transplantation
  Arms: autologous mitochondria transplantation
Drug: intracytoplasmic sperm injection (ICSI) — intracytoplasmic sperm injection (ICSI)
  Arms: ICSI

SUMMARY:
Embryo quality was ranked as one of the most important predictors in determining the success of implantation, while clinically some patients may experience repeated IVF failure due to persistent poor embryo quality.Mitochondria, as the energy factory, is confirmed being a hallmark of quality and developmental potential of human oocytes, and decreased mitochondria copy number was reported to be associated with oocyte aging and dysfunctional mitochondria would be expected to influence the late stages of oocyte maturation and early embryogenesis.The objective of this study is to evaluate the effect of mitochondria transfer from bone marrow mesenchymal stem cell on the quality of oocyte.

DETAILED DESCRIPTION:
This study is a pilot study to investigate the effect of autologous mitochondria transplantation for improving oocyte quality.

Design: randomized controlled trial. Setting: Assisted reproductive technologies unit. Patients: patients who is in accordance with the inclusion criteria, and not meet the exclusion criteria, who had repeated IVF treatment from Sep 2018 to Sep 2021.

Intervention: The comparison was made between mitochondria transfer（MIT) group and the control group, both groups are conducted with the GnRH-a super-long protocol for IVF treatment. MIT group injects autologous mitochondria from bone mesenchymal stem cells into oocyte.

Main outcome measures: The primary outcome of the study is live birth rate. The secondary outcomes were clinical pregnancy rate, number of oocytes retrieved, fertility rate, normal fertilization rate, rate of transferable embryo and good quality embryo rate.

ELIGIBILITY:
Inclusion Criteria:

1. Women age >20 years and <43 years.
2. Anti-müllerian hormone（AMH） level ≥1.1 ng/ml.
3. Previous failed transfer cycle ≥2.
4. BMI>18kg/m2 and <25kg/m2.
5. Written informed consent.

Exclusion Criteria:

1. Abnormal uterine development, endometrial adhesion or previous endometrial dysplasia (<7mm)
2. Other medical diseases that cannot be pregnant.
3. Complicated with adenomyosis, endometriosis confirmed by surgery, ovarian endometriosis cyst ≥2 cm by ultrasound, all kind of malignant tumors or precancerous disease.
4. Untreated hydrosalpinx.
5. The man has definite factors that affect the quality of the embryo, such as persistent abnormal DNA fragment rate (>30%) and non-obstructive spermatozoa.
6. Intracytoplasmic sperm injection with donor.

Eliminate or falls off Criteria:

1.The number of retrieved oocytes <6.

Ages: 20 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
live birth rate | 2-3years
  number of live birth/ transferred cycle.Compare the live birth rate between the two groups with SPSS 20.0.

SECONDARY OUTCOMES:
clinical pregnancy rate | 2-3years
  Clinical pregnancy means pregnancy sac is seen intrauterine under ultrasound 7 weeks after embryo transferred.
  Clinical pregnancy rate(%): number of clinical pregnancy/transferred cycle.Compare the clinical pregnancy rate between the two group with SPSS 20.0.
number of oocytes retrieved | 2-3years
  Compare the number of oocytes retrieved between the two group with SPSS 20.0.
fertility rate | 2-3years
  Fertility rate(%): number of oocyte fertilized/ number of oocytes retrieved.Compare the fertility rate between the two group with SPSS 20.0.
normal fertility rate | 2-3years
  Normal fertility rate(%): number of oocyte normally fertilized/ number of oocytes retrieved. Compare the normal fertility rate between the two group with SPSS 20.0.
good quality embryo rate | 2-3years
  Cleavage embryo grades 1 or 2 with 6-10 blastomeres were considered good quality embryos. Good quality embryo rate(%): number of good quality embryo/number of fertilized oocytes.Compare the good quality embryo rate between the two group with SPSS 20.0.